CLINICAL TRIAL: NCT03910166
Title: Prospective, Multi-center and Randomized Controlled Clinical Study to Verify Effectiveness and Safety of Drug-eluting Balloon in PTA Procedure of Vertebral Artery Ostium Stenosis
Brief Title: AcoArt VI / Vertebral Artery Ostium Stenosis in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acotec Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acotec-06
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-01

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: drug eluting balloon catheter; stenting
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB group (Experimental): use DEB catheter(trade name:Orchid/Dhalia) to treat the stenosis or occlusion in Vertebral Artery Ostium Stenosis of experimental arm
  Interventions: Procedure: drug-coated balloon catheter（Orchid, Acotec）
- BMS group (Active Comparator): use Intracranial artery stent system(trade name:Apollo) to treat stenosis or occlusion in Vertebral Artery Ostium Stenosis of control group
  Interventions: Procedure: Intracranial artery stent system（APOLLO）

INTERVENTIONS:
Procedure: drug-coated balloon catheter（Orchid, Acotec） — After predilation, using drug-coated balloon catheter to cover the whole treated segment
  Arms: DCB group
Procedure: Intracranial artery stent system（APOLLO） — stent assisted angioplasty
  Arms: BMS group

SUMMARY:
The purpose of this study is to determine whether DEB is not inferior to common bare metal stent using under in long-term vessel patency and inhibiting restenosis in Vertebral Artery Ostium Stenosis

DETAILED DESCRIPTION:
Vertebral Artery Origin Stenting is an established alternative to open surgical bypass for the treatment of Vertebral Artery Ostium Stenosis .

DEBs are designed to promote arterial patency by reducing neointimal proliferation.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 80 years old
* symptomatic VAO stenosis refractory to AMM (aggressive medical management)
* etiology of VAOS was atherosclerosis
* the diameter of the normal segment of the artery beyond the stenosis between 3mm and 5mm
* Target lesion has stenosis ≥ 70% evidenced by angiography
* Score on the modified Rankin scale ≤ 3
* NIHSS≤ 6
* Patients have signed informed consent

Exclusion Criteria:

* In-stent restenosis in vertebral artery
* Severe calcified lesion or residual stenosis ≥30% after predilatation or flow-limiting dissection
* Tortuous or variable vessels
* distal serial stenosis or distal vascular dysplasia of the stenosis segment
* Non-atherosclerotic arterial stenosis
* Non-vertebral artery stenosis caused TIA or stroke
* intracranial stent implantation within 12 months
* Intracranial hemorrhage occurred within 3 months
* Obvious thrombosis in brain vessel, or have received thrombolytic therapy 24 hours before procedure
* Active bleeding or coagulation disorders
* Serious liver/kidney damage, not suitable for routine surgical treatment
* Myocardial infarction or extensive cerebral infarction occurred within 2 weeks
* Uncontrolled high blood pressure
* Complicated intracranial tumor, cerebral arteriovenous malformation, or intracranial aneurysm
* Potential sources of cardiogenic thrombosis, such as mitral stenosis, atrial septal defect, aorta or mitral valve replacement, left atrial myxoma, etc
* Life expectancy shorter than 1 years
* Patients whit cognitive impairment or mental disorders
* Known hypersensitivity to aspirin, heparin, clopidogrel,paclitaxel, contrast medium, etc
* Pregnant and lactating women
* Patients who have participated in other clinical trials during the same period that lead to researchers who believe that patients may not be able to follow the trial program

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of target lesion restenosis | 12Months
  Target Lesion Restenosis（diameter stenosis ≥50%） under DSA at 12 Months or diamater stenosis ≥50% under DSA before Target Lesion Revascularization within 12 Months
Rate of device success | during the operation
  DEB group: DEB catheter can reach the target lesions, expand as expected (not broken),and withdraw successfully. BES group: the stenosis rate of proximal outflow less than 50% with intervention and no ischemia or hemorrhage occurred.

SECONDARY OUTCOMES:
Rate of device success | during the operation
  DEB group: DEB catheter can reach the target lesions, expand as expected (not broken),and withdraw successfully. BES group: the stenosis rate of proximal outflow less than 50% with intervention and no ischemia or hemorrhage occurred.
Incidence of hemorrhagic stroke and posterior circulation ischemic stroke | 12 Months
  incidence of hemorrhagic stroke and posterior circulation ischemic stroke within 12 months
Incidence of transient ischemic attack of posterior circulation | 12 Months
  incidence of transient ischemic attack of posterior circulation within 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Jiao, PhD, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu hospital, Beijing, China

REFERENCES:
- [Derived] Luo J, Jiang C, Wang H, Peng R, Wang T, Kuai D, Liang G, Wang F, Wang S, Xu C, Chen W, Deng J, Hu X, Wan S, Li B, Yin B, Du Y, Cheng G, Wan J, Chen X, Wang Y, Jiao L; DCB-VAOS Trial Investigators. Effect of drug-coated balloon in patients with severe vertebral artery origin stenosis: A multicenter randomized controlled trial. Int J Stroke. 2025 Oct 9:17474930251377055. doi: 10.1177/17474930251377055. Online ahead of print. PMID 41067866
- [Derived] Wang Y, Ma Y, Gao P, Chen Y, Yang B, Feng Y, Jiao L. Paclitaxel Coated Balloon vs. Bare Metal Stent for Endovascular Treatment of Symptomatic Vertebral Artery Origin Stenosis Patients: Protocol for a Randomized Controlled Trial. Front Neurol. 2021 Jan 18;11:579238. doi: 10.3389/fneur.2020.579238. eCollection 2020. PMID 33584491